CLINICAL TRIAL: NCT02422147
Title: Endoscopic Ultrasound (EUS)-Guided Ablation of Pancreatic Cyst Neoplasms
Brief Title: EUS-guided Ablation of Pancreatic Cyst Neoplasms
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 723324
Record Dates: First submitted 2015-02-24; First posted 2015-04-21 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ablation of PCL: Patients with pancreatic cysts will undergo ablation using alcohol under EUS-guidance
  Interventions: Procedure: Ablation of PCL

INTERVENTIONS:
Procedure: Ablation of PCL — All procedures are standard of care and will be undertaken using a curvilinear echoendoscope. The cyst will be punctured using a 22G needle and after subtotal evacuation of the cyst, injection is performed with a volume of alcohol that is equal to the quantity aspirated, and the cyst will be lavaged for 3 to 5 minutes. The injected ethanol will then be evacuated at the end of lavage, leaving just enough fluid to outline the cavity. A second ablative agent such as paclitaxel is then injected and left in the cyst cavity. At the completion of the procedure, the needle will be removed from the cyst cavity.
  Other Names: EUS-guided ablation of pancreatic cyst lesions (PCL)

SUMMARY:
This is a registry that will maintain prospective data on the clinical outcomes of all patients with pancreatic cyst lesions who undergo EUS-guided alcohol ablation.

DETAILED DESCRIPTION:
Visit 1 for all participants will consist of going over the Informed Consent form and talking with the patient about the study. If the patient agrees to participate, he/she will be asked to sign the form, and a copy will be given to him/her for his/her records. This will be conducted during the day of the endoscopic procedure before the participant is under anesthesia. The treatment provided will be standard-of-care that is offered to patients with pancreatic cyst lesions (PCL) interested in undergoing EUS-guided ethanol ablation.

An MRI of the abdomen will be obtained as baseline measure to determine the size of the pancreatic cyst and confirm diagnosis.

Prior to undertaking any ablation, the cyst fluid will be sampled at a prior EUS session to check for mucin, viscosity, carcinoembryonic antigen (CEA) (>200U/L=mucinous cyst), amylase and if required molecular marker analysis. Once a PCL is determined to have a malignant potential the patient will be selected for EUS-guided ablation. All patients will receive a dose of intravenous ciprofloxacin 500mg 30 minutes prior to the ablation. These evaluation and treatment measures are standard-of-care for any patient with pancreatic cyst lesion undergoing EUS-guided ethanol ablation.

Procedural Technique: All procedures will be undertaken using a curvilinear echoendoscope. Once a cyst is identified for ablation it will be punctured using a 22G needle. After subtotal evacuation of the cyst, injection is performed with a volume of alcohol that is equal to the quantity aspirated, and the cyst will be lavaged for 3 to 5 minutes, alternatively filling and emptying the cavity. The injected ethanol will then be evacuated at the end of lavage, leaving just enough fluid to outline the cavity. A second ablative agent such as paclitaxel is then injected and left in the cyst cavity; the volume injected should not exceed the volume of aspirated fluid. The needle tip must be carefully maintained within the cyst to avoid parenchymal injury or cyst wall leak. At the completion of the procedure, the needle will be removed from the cyst cavity. When a cyst is not restored to its original size during ethanol injection, vigorous lavage and aspiration must be avoided because of probable communication with the main pancreatic duct.

In patients with multi-loculated cysts, a single injection may not provide sufficient drug delivery to all locules within a cyst. It is important to determine the optimal angle at which the needle can be introduced into the maximum number of targeted locules. When all punctured locules cannot be visualized on endosonographic image, needle passage across a septation may be indicated. The simultaneous collapse of locules across the septum during cyst fluid evacuation and spread of echogenic bubbles across the septation during injection of ablative agents are indication of good distribution of the ablative agent into the locules. This is important as a missed locule may result in cyst regrowth and treatment failure. While additional needle passes through different angles may increase the effectiveness of cyst ablation it will also increase the incidence of adverse events. Therefore a second needle puncture may be considered only when the risk of adverse events appears low.

The relative effectiveness of the procedure is related to the degree of contact between the ablative agent and the cyst epithelium. However, it is important to maintain the needle in the visual plane and within the cyst cavity during the entire procedure. All techniques described above are standard-of-care treatment measures offered to patients undergoing EUS-guided ethanol ablation of pancreatic cysts.

Ablative agents:

1. Ethanol: concentration of 80-99% may be used.
2. Paclitaxel: Because of the high viscosity of its cosolvent (castor oil) the paclitaxel solution must be diluted 1:1 in 0.9% normal saline to yield a final dose concentration of 3mg/mL. However, if the agent is available in a less viscous format (polymeric micelle) it can be used without dilution (a dose concentration of 6mg/mL).

Follow-up:

1. Patients will be admitted overnight for observation and kept nil by mouth. A complete blood count and serum amylase level will be checked the next day and patients will be discharged home if clinically well, with no evidence of pancreatitis or other adverse events and can tolerate a low fat diet. Patients will be prescribed oral ciprofloxacin 500 mg to be taken twice a day for three days. This will be standard-of-care follow-up.
2. A CT of the abdomen will be obtained at 3 months to assess treatment response. If there is no change in size of the cyst, further CT scans will be scheduled at 3-month intervals with another attempt at EUS-guided cyst ablation. If there is complete or partial cyst resolution, follow-up CT scans will be obtained at 6-month intervals. If complete resolution is documented on two CT scans, then the patient will be scheduled for annual CT scans. This will be standard-of-care follow-up. 3. Patients with persistent or only partial cyst resolution despite two ablative treatment sessions will be referred to a pancreatic surgeon for consultation. If the patients are high-risk surgical candidates, surveillance by EUS and cross-sectional imaging will be continued per International Society of Pancreatology guidelines. This will be standard-of-care follow-up. 4. Definitions: Using multi-detector CT scans and specialized software the original volume (OV) of the cyst will be calculated by the radiologist. Complete resolution will be defined as the cyst being nonvisible or less than 5% of the OV on follow-up CT; Partial resolution of the cyst will be defined as decrease in size by 5-25% of the OV and the cyst will be defined as Persistent if > 25% the OV.

ELIGIBILITY:
Inclusion Criteria:

1. Benign branch-duct intraductal papillary mucinous neoplasm (IPMN) or mucinous cyst neoplasm (MCN) measuring >2 and up to 4cm in size and located in the head or body of the pancreas.
2. Benign branch-duct IPMN or MCN measuring > 2 and up to 4cm in size and located in the tail of the pancreas in a high-risk surgical candidate.
3. A branch-duct IPMN or MCN with high-risk features (mural nodule or enlarging in size) in a high-risk surgical patient.
4. Indeterminate cyst lesions

Exclusion Criteria:

1. Cysts measuring <2cm or >4cm.
2. Multiloculated cysts (>4 locules).
3. Cysts with vascular supply.
4. Cysts communicating with the main pancreatic duct via an obvious side-branch measuring 2mm or more in diameter.
5. Cysts with hypoechoic mass lesions that on fine needle aspiration (FNA)reveal malignant cells.
6. Recent history of pancreatitis and EUS findings suggestive of a pseudocyst.
7. Bleeding tendency; international normalized ratio (INR) >1.4 or platelet count <70,000.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any male or female presenting to Florida Hospital Center for Interventional Endoscopy with a pancreatic cyst will be considered for this registry pending he/she meets inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
This study will evaluate the clinical outcomes (effectiveness) of all patients with pancreatic cyst lesions undergoing EUS-guided ethanol ablation. This will include complete resolution of the pancreatic cyst lesion at the end of the treatment period. | Up to 12 months
  Clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript will be developed and submitted for publication upon study completion.